CLINICAL TRIAL: NCT05335980
Title: A Phase II Prospective, Single-Arm, Open-Label, Multi-Center Study Using the Nu-V3 Cranial Nerve Stimulation Treatment Device in Patients With Chronic Pain, Anxiety, Depression, and/or Sleeplessness
Brief Title: Nu-V3 Non-Invasive Nerve Stimulation Device Trial for Chronic Pain, Anxiety, Depression, Sleeplessness
Acronym: Nu-V3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Nu-Life Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nu-V3 CPADS PROTOCOL
Record Dates: First submitted 2018-03-28; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pain; Anxiety; Depression; Sleeplessness
Keywords: Device; TENS; Neuromodulation; PTSD; Neuropathy; Inflammatory; Arthritis; Chronic Pain; Fibromyalgia; Osteoarthritis; TMJ; Insomnia
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic; Arthritis; Fibromyalgia; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: A Phase II Prospective, Single-Arm, Open-Label, Multi-Center Study Using the Nu-V3 Cranial Nerve Stimulation Treatment Device in Patients with Chronic Pain, Anxiety, Depression, and/or Sleeplessness
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Nu-V3 Device (Experimental): Treatment with the Nu-V3 Device.
  Interventions: Device: Nu-V3

INTERVENTIONS:
Device: Nu-V3 — The Nu-V3 device provides a continuous flow of intermittent, low frequency electrical pulses to the ear's specific cranial nerve endings. This treatment is delivered 24 hours a day for the first 12 weeks, then is delivered two weeks on, one week off for the following 12 weeks.

SUMMARY:
The Nu-V3 Clinical Study is a prospective, single-arm, open-label, multi-center study using the Nu-V3 cranial nerve stimulation treatment device in patients with chronic pain, anxiety, depression, and/or sleeplessness.

For this Phase II study, a total of 100-200 patients at multiple centers will be registered for study participation. Study participants are those who have signed the informed consent form, met the inclusion and exclusion criteria, and are enrolled in the study at one of multiple sites. Enrolled participants are stratified based on their chronic pain, anxiety, depression, and/or sleeplessness symptom presentation at baseline and treated with the Nu-V3 device for 24 weeks. Interim analysis of reported data will be based on baseline stratifications and conducted at 6, 12, 18, and 24 weeks during this time. The participant will be evaluated after the initial 12-week treatment period to assess for further therapeutic need. Upon having three consecutive weeks of mean symptom reduction of ≥70% via patient reported numerical scales, the participant will continue as described in the study assessments table, but without device therapy. Then if the participant's primary symptom score increases at any time by ≥20%, they may again continue device therapy until week 24.

DETAILED DESCRIPTION:
Subjects enrolled onto the Nu-V3 Clinical Trial will undergo the following regimen:

* At the baseline visit, patients will be asked to complete study questionnaires regarding all of the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their quality of life, active medications, medical history, and demographic information. The subject's primary symptom of concern will also be notated at baseline, for later assessment of continuation after week 12.
* At each subsequent visit, patients will be asked to complete study questionnaires regarding all the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their activity level and quality of life.
* The sessions will begin with the Nu-V3 device being clipped on the ear and three small pads (non-invasive) adhered to the surface of the ear. Each Nu-V3 device lasts for up to 14 days with a change in the pads approximately 7 days into the treatment.
* Each session takes approximately 15-20 minutes. The placement of the device takes approximately 5 minutes and the remaining time is spent verifying ePRO form completion, and evaluating the patient for all device effects.
* The Nu-V3 device is mobile and is worn externally on the left ear 24 hours a day during treatment, fitting comfortably behind the ear. An electrical signal is sent to the external ear through coated wire leads attached to the device and adhesive pads which attach to three sites on the ear.
* Participants should be able to perform their typical day-to-day activities while wearing the device. They may shower while wearing the Nu-V3 device, provided that they do not get the device wet and use the small disposable ear covers that are provided for them.
* In the event the Nu-V3 gel pads are inadvertently removed or the device comes off, the participant will contact the site coordinator. The participant is encouraged to adjust the device placement as needed for comfort.
* Patients should not change their existing forms of treatment or medications without discussion with the study investigator.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years of age
* Participant presents with one or more of the following symptoms: pain, depression, anxiety, and/or sleeplessness
* Participant is capable of understanding the use and maintenance of the device
* Participant is capable and agreeing to participate in the ongoing assessment
* Participant has signed the Informed Consent Form
* Participant can commit to follow all protocol study timepoints

Exclusion Criteria:

* Participants with a Pacemaker
* Participants with irregular heart rate or a heart rate lower than 60 beats per minute (bradycardia)
* Have had a transplant within the last 2 years
* Have had a heart attack or cardiac bypass surgery within the last 12 months
* History of substance abuse, including prescription drugs, within the last 12 months
* Patients with complaints of dizziness or lightheadedness within the last 3 months
* Women who are pregnant
* Participants with Diabetic Retinopathy
* Current Ear infection
* SBP < 100 and/or DBP < 60
* History of uncontrolled bipolar disorder within the last 12 months
* History of uncontrolled seizures within the last 12 months
* History of Aneurysms
* History of syncope within the last 12 months
* Participants that have had a TIA or stroke within the last 12 months
* Participants with health problems deemed at risk for the study by the Principal Investigator
* Participants with any changes to Pain/Anxiety/Depression/Sleeplessness medications within last 60 days (participants that do not meet this medication- change washout period may be delayed until 60-day period is met)
* Participants that are currently under adjudication process for disability support, VA or other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness and overall change in reported primary symptom of concern: Chronic Pain | 12 and 24 weeks
  Chronic Pain - (PEG Scale) The PEG is a three-item instrument that measures pain intensity (one item) and pain interference (two items). The PEG is a three-item instrument that measures pain intensity (one item) and pain interference (two items). Each item is valued from 0 (no pain/interference) to 10 (as bad as you can imagine). The instrument score is calculated as the average of the three item values.
Effectiveness and overall change in reported primary symptom of concern: Anxiety | 12 and 24 weeks
  Anxiety - (GAD-7)The GAD-7 is a seven-item instrument that measures respondents' symptoms of anxiety. The GAD-7 is a seven-item instrument that measures respondents' symptoms of anxiety. Each item is scored on a four-point Likert scale, and values range from 0 ("Not at all") to 3 ("Nearly every day".) Items are summed to determine the instrument's score. Values of 10 or higher have been associated with moderate anxiety, while values of 15 or higher have been associated with severe anxiety.
Effectiveness and overall change in reported primary symptom of concern: Depression | 12 and 24 weeks
  Depression - (PHQ-9) The PHQ-9 is a nine-item instrument that measures depression-related symptoms and functional impairment. The PHQ-9 is a nine-item instrument that measures depression-related symptoms and functional impairment. Each item is scored on a four-point Likert scale and values range from 0 ("Not bothered at all") to 3 ("Bothered nearly every day.") The items' values are summed to determine the instrument's score. PHQ-9 values of 10 and 15 represent moderate and moderately severe depression respectively.
Effectiveness and overall change in reported primary symptom of concern: Sleeplessness | 12 and 24 weeks
  Sleeplessness - PROMIS short form 4a- This eight item instrument measures sleep disturbance and sleep-related impairment. This eight item instrument measures sleep disturbance and sleep-related impairment.

SECONDARY OUTCOMES:
Effectiveness: Symptom Frequency | 12 and 24 weeks
  In the Nu-V3 device treatment arm, the study will report the mean time from treatment initiation to reduction of symptoms of at least 30% in any of the four domains of symptom measurement.
Effectiveness: Symptom Severity | 12 and 24 weeks
  In both the Nu-V3 device treatment arm and the observation arm, the study will report the mean percentage change in symptoms severity from initiation to 12 and 24 weeks for each instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Doebbeling, MD, Study Chair — Nu-Life Solutions; Kamran Chaudhary, MD, Principal Investigator — Nu-Life Solutions; Eric T Siebeneck, MS, Study Director — Nu-Life Solutions
Locations (1):
- Arizona Endocrinology, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Nu-Life Solutions Homepage — https://www.nu-v3.com/

DOCUMENTS (3):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT05335980/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT05335980/SAP_001.pdf
  • Informed Consent Form (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT05335980/ICF_002.pdf